CLINICAL TRIAL: NCT06249685
Title: Does Wearing Hearing Aids Impact the Affective State of Older Adults With Hearing Loss in Their Daily Lives?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO-FY2020-252
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Emotions; Stress Physiology
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: ABA Repeated Reversal design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Baseline-Unaided (No Intervention): No hearing aids.
- Aided (Experimental): Fitted with bilateral hearing devices.
  Interventions: Device: Bilateral hearing devices
- Follow-up-Unaided (No Intervention): No hearing aids.

INTERVENTIONS:
Device: Bilateral hearing devices — Three week trial while wearing bilateral hearing devices.
  Other Names: Hearing aid; Hearing aids; Receiver-in-the-canal; RIC
  Arms: Aided

SUMMARY:
The proposed field trial will clarify the real-world effectiveness of HAs in remediating deficits in emotion processing for older adults with mild-to-moderate hearing loss. This study will employ a repeated reversal design to establish baseline affective state without HAs, when wearing amplification, and after HAs are removed. This study will triangulate self-report, behavioral, and physiological measures to capture nuances of emotional processing in the laboratory and in daily listening. Naturalistic stimuli will be used as it occurs in daily life to elicit emotional experiences, and ecological momentary assessment and commercially-available wearable sensors will be used to track changes in emotional state in daily listening. Anchoring real-world emotional experiences with controlled laboratory experiences will validate wearable sensors. Additionally, laboratory emotional stimuli will be related to real-world emotional experiences to establish the utility of laboratory stimuli in future studies. It is likely that benefits in emotional processing will have differential effects based on individual characteristics (such as degree of hearing loss, age, gender, cognitive ability, and personality), so participants will be analyzed according to larger groupings based on individual differences.

DETAILED DESCRIPTION:
Thirty-five participants will complete preliminary measures, including assessments of routine audiometrics, demographics, personality, and working memory. For each arm of the trial (baseline-unaided; aided; follow-up unaided) participants will be issued sensors to use while pursuing normal daily life activities. These sensors can provide information such as heart rate (HR) and respiration activity, which have been associated with the arousal dimension of emotion. Participants also will download a mobile app that will automatically prompt them throughout their day to indicate their perceived arousal and valence and listening-related workload. For each arm of the trial interindividual and intraindividual emotion perception, speech understanding, and perceived workload will be also be assessed using laboratory-based self-report, behavioral, and physiological measures. Subjective measures of hearing aid benefit, emotional consequences of hearing loss, and the effect of hearing loss on emotional communication will be assessed through validated questionnaires at the conclusion of each arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral, uncomplicated, adult-onset mild-to-moderate hearing loss.
* No previous experience with hearing aids
* Fluent English speakers
* Have adequate literacy and cognitive competence to complete informed consent and required questionnaires with minimal assistance.
* Able to transport themselves to the data collection site and participate in the study without assistance from researchers.

Exclusion Criteria:

* History of otologic surgery or chronic middle or outer ear pathology
* Evidence of retrocochlear involvement
* Known psychiatric or neurologic disorder.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Self-reported arousal | Measured several times per day for 6 days in each arm of the study (ecological momentary assessment); and at a lab appointment on day 7; day 28; and day 35 of the trial.
  Arousal rating measured with the Self-assessment manikin (SAM)
Self-reported valence | Measured several times per day for 6 days in each arm of the study (ecological momentary assessment) and at a lab appointment on day 7; day 28; and day 35 of the trial.
  Valence rating measured with the Self-assessment manikin (SAM)

SECONDARY OUTCOMES:
Self-reported task-load | Measured several times per day for 6 days in each arm of the study (ecological momentary assessment) and at a lab appointment on day 7; day 28; and day 35 of the trial.
  Task-load rating measured with the NASA-TLX
Physiological arousal - heart rate | easured several times per day for 6 days in each arm of the study (ecological momentary assessment) and at a lab appointment on day 7; day 28; and day 35 of the trial.
  Heartbeats per minute
Physiological arousal - respiration activity | easured several times per day for 6 days in each arm of the study (ecological momentary assessment) and at a lab appointment on day 7; day 28; and day 35 of the trial.
  Breaths per minute
Physiological arousal - electrodermal responses | Day 7; day 28; and day 35 of the trial.
  Skin conductance in response to emotionally evocative sounds (International Affective Digital Sounds) at soft, average, loud levels
Physiological valence - electromyography | Day 7; day 28; and day 35 of the trial.
  Facial sEMG in response to emotionally evocative sounds (International Affective Digital Sounds) at soft, average, loud levels
Emotion identification - Toronto Emotional Speech Set | Day 7; day 28; and day 35 of the trial.
  Percent correct identification of emotion contained in auditory stimuli at soft, average, loud levels
Word recognition - Toronto Emotional Speech Set | Day 7; day 28; and day 35 of the trial.
  Percent correctly identified single word auditory stimuli at soft, average, loud levels
Abbreviated Profile of Hearing Aid Benefit (APHAB) | Day 7; day 28; and day 35 of the trial.
  Validated questionnaire that assesses frequency of problems with speech communication and aversiveness of sounds in daily listening
Hearing Handicap Inventory for Elderly-Screening version (HHIE-S) | Day 7; day 28; and day 35 of the trial.
  Validated questionnaire that measures the effects of hearing impairment on emotional and social adjustment
Emotional Communication in Hearing Questionnaire (EMO-CHeQ) | Day 7; day 28; and day 35 of the trial.
  Validated questionnaire that assesses benefits of hearing aids in addressing emotional communication.

CONTACTS AND LOCATIONS:
Overall Officials: Jani A Johnson, PhD, Principal Investigator — University of Memphis
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No